CLINICAL TRIAL: NCT02345980
Title: A Randomized Controlled Trial Evaluating Sildenafil Citrate in Relieving Ureteral Stent Related Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed R. EL-Nahas, Urology & Nephrology Center, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sildenafil and USS
Record Dates: First submitted 2014-10-01; First posted 2015-01-26 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Quality of Life
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Active Comparator): Patient in this arm will receive sildenafil citrate 50 mg tablet once daily after ureteral stent fixation.
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): Patient in this arm will receive placebo daily after ureteral stent fixation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil
  Other Names: Viagra
  Arms: Sildenafil
Drug: Placebo
  Arms: Placebo

SUMMARY:
Despite its beneficial effect, ureteral stents may produce symptoms (such as hematuria, dysuria, frequency, urgency, urge incontinence and suprapubic or flank pain) that affect the quality of life in 70-80%.

This study will be conducted to evaluate the role of Phosphodiestrase 5 inhibitor (Sildenafil Citrate) in relieving these symptoms.

DETAILED DESCRIPTION:
Adult patient (>18 years) who will undergo ureteral stent fixation after endoscopic procedures will be randomized between the study arms.

Exclusion criteria:

1. Patients who had lower urinary tract symptoms before stent fixation.
2. Ureteral stent fixation after open surgery.
3. Known contraindications to Sildenafil Citrate

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged >18 years

Exclusion Criteria:

1. Patients who had LUTS before DJ stent fixation
2. DJ stent fixation after open surgery
3. Contraindication to Sildenafil citrate

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Ureteral Stent Symptoms Questionnaire (USSQ) Score | 2-4 weeks
  Comparison of total USSQ scores between study arms.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 2-4 weeks
  Analyzing frequency and severity of side effects of Sildenafil

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed R EL-Nahas, MD, Principal Investigator — Urology and Nephrology Center, Mansoura University, Egypt
Locations (1):
- Urology and Nephrology Center, Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Derived] Tharwat M, Elsaadany MM, Lashin AM, El-Nahas AR. A randomized controlled trial evaluating sildenafil citrate in relieving ureteral stent-related symptoms. World J Urol. 2018 Nov;36(11):1877-1881. doi: 10.1007/s00345-018-2339-y. Epub 2018 May 15. PMID 29766318